CLINICAL TRIAL: NCT07099547
Title: A Study to Evaluate the Efficacy and Safety of ZG005 in Combination With Platinum-Based Chemotherapy as First-Line Treatment in Participants With Advanced Biliary Tract Carcinoma
Brief Title: Study of ZG005 in Combination With Platinum-Based Chemotherapy in Participants With Advanced Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-007
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text group (Experimental): ZG005+Gemcitabine +Cisplatin
  Interventions: Drug: ZG005; Drug: Gemcitabine; Drug: Cisplatin
- Control group (Experimental): Tislelizumab+Gemcitabine+Cisplatin
  Interventions: Drug: Tislelizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: ZG005 — ZG005 20 mg/kg IV Q3W
  Arms: Text group
Drug: Tislelizumab — Tislelizumab 200mg IV Q3W
  Arms: Control group
Drug: Gemcitabine — Gemcitabine 1000mg/m^2 Q3W. Gemcitabine will be administered on D1/D8 in every three weeks cycle.
Drug: Cisplatin — Cisplatin 25mg/m^2 Q3W. Cisplatin will be administered on D1/D8 in every three weeks cycle.

SUMMARY:
This is a randomized, open-label, phase II study evaluating first-line treatment for advanced gallbladder cancer. It aims to assess the efficacy, safety, pharmacokinetics, and immunogenicity of the ZG005 in Combination with gemcitabine and cisplatin as first-line therapy in Participants with advanced gallbladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Subjects with a histopathological or cytologically diagnosis of Gallbladder cancer.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Participants were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China